CLINICAL TRIAL: NCT00208637
Title: He Purongo Mo Nga Kai Hei Arai i Te Matehuka - Dietary Diabetes Prevention Study for Maori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edgar National Centre for Diabetes Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kai Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Insulin Resistance
Keywords: Maori; insulin sensitivity; cardiovascular risk; diabetes prevention; diet modification
MeSH Terms: conditions — Insulin Resistance | interventions — Diet, High-Protein; Diet

INTERVENTIONS:
Behavioral: moderate carbohydrate, high protein diet (MCHP)
Behavioral: high carbohydrate-high fibre (HCHF) diet

SUMMARY:
High protein diets are popular among Maori, especially on the East Coast of the North Island. The purpose of this study was to compare the metabolic effects of a moderate carbohydrate, high protein diet (MCHP) with a high carbohydrate-high fibre (HCHF) diet on insulin sensitivity in Maori at increased risk of developing diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
This was a 6-month pilot intervention study of self-identifying Maori participants in a randomised control trial conducted in Dunedin and Invercargill. The study consisted of three, two month phases and was conducted over a period of six months. Participants meeting all the inclusion criteria were randomised into three groups: moderate carbohydrate-high protein (MCHP), high carbohydrate-high fibre (HCHF) or a control group. Those randomised to the experimental diets were recommended an energy intake based on their current BMI levels. The aim of phase one was to achieve weight loss with weekly advice and support from the research team. The aim of phase two was for weight maintenance with continued weekly advice and support. Phase three consisted of a weight maintenance phase without support. Those in the control group were instructed to follow their own self selected diet plan.

Outcome was determined by examining surrogate clinical endpoints. The clinical endpoints included the following recorded measurements of anthropometric measurements, bioelectrical impedance measurements, profile of mood state questionnaires, activity questionnaires, and three day diet records were collected at 0, 2, 4 and 6 month periods. Biochemical measures of lipid profile, fasting insulin and glucose, liver functions and uric acid levels were also conducted.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Maori aged between 17-75 years
* Male and female
* Non-diabetic
* Resident of Dunedin and Invercargill
* BMI >27
* Family history of T2D

Exclusion Criteria:

* The presence of diabetes, renal or liver failure, or any other medical condition which is unstable and for which potential partcipants are currently having active treatment.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2002-08; Study Completion 2004-12

PRIMARY OUTCOMES:
Dietary intake as measured by 3-day weight diet records

SECONDARY OUTCOMES:
Blood pressure
Bioelectric Impedence
Weight
Waist circumference
Total cholesterol and lipid subfractions (LDL, HDL)
Fasting insulin
Lipoprotein A + B
Inflammatory markers
Urinary albumin:creatinine ratio
Quality of life
All measures to be compared at end of study (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Brooking, BSc, MA, Principal Investigator — Edgar National Centre for Diabetes Research, Dunedin, NZ; Jim I Mann, FRACP, PhD, Study Director — Edgar National Centre for Diabetes Research, Dunedin, NZ
Locations (1):
- Edgar National Centre for Diabetes Research, Dunedin, Otago, New Zealand

REFERENCES:
- [Derived] Brooking LA, Williams SM, Mann JI. Effects of macronutrient composition of the diet on body fat in indigenous people at high risk of type 2 diabetes. Diabetes Res Clin Pract. 2012 Apr;96(1):40-6. doi: 10.1016/j.diabres.2011.11.021. Epub 2011 Dec 16. PMID 22178004
- See also: Edgar National Centre for Diabetes Research, NZ website — http://www.otago.ac.nz/diabetes